CLINICAL TRIAL: NCT00003497
Title: Phase II Study of Antineoplastons A10 and AS2-1 Capsules In Patients With Non Small Cell Lung Cancer
Brief Title: Antineoplaston Therapy in Treating Patients With Stage IV Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066536; BC-LA-10 (Other: Burzynski Research Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Stage IV Non-small Cell Lung Cancer
Keywords: recurrent non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antineoplastons (Experimental): Antineoplaston therapy (Atengenal + Astugenal) capsules orally six to seven times a day. Treatment continues in the absence of disease progression or unacceptable toxicity. absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Antineoplaston therapy (Atengenal + Astugenal) capsules orally six to seven times a day. Treatment continues in the absence of disease progression or unacceptable toxicity. absence of disease progression or unacceptable toxicity.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
Current therapies for Stage IV non-small cell lung cancer provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of Stage IV lung cancer

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on patients with Stage IV lung cancer.

DETAILED DESCRIPTION:
Stage IV non-small cell lung cancers receive Antineoplaston A10 and AS2-1 capsules orally six to seven times a day. Treatment continues in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with Stage IV non-small cell lung cancer, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with Stage IV non-small cell lung cancer.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 4 months for 2 years, every 6 months for 2 years, and then annually for 2 years thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV non-small cell lung cancer that cannot be cured with existing therapeutic regimens
* Measurable disease by CT scan or MRI

  * Tumor must be at least 2 cm for the lymph nodes located in the head, neck, axillary, inguinal or femoral areas and at least 0.5 cm for other areas

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* No hepatic insufficiency
* Bilirubin no greater than 2.5 mg/dL
* SGOT and SGPT no greater than 5 times upper limit of normal

Renal:

* No renal insufficiency
* Creatinine no greater than 2.5 mg/dL

Cardiovascular:

* No chronic heart failure
* No uncontrolled hypertension

Pulmonary:

* No serious lung disease (e.g., severe chronic obstructive pulmonary disease)

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No other serious medical or psychiatric conditions
* No active infection
* No serious malabsorption syndromes

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* At least 8 weeks since prior radiotherapy (less than 8 weeks if multiple tumors are involved) and recovered

Surgery:

* No prior extensive stomach or intestinal surgery
* Recovered from any prior surgery

Other:

* Prior cytodifferentiating agents allowed
* No prior antineoplaston treatment
* No other concurrent treatment for metastatic lung cancer

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 1996-08-21 (Actual); Primary Completion 1998-02-02 (Actual); Study Completion 1998-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com